CLINICAL TRIAL: NCT01696903
Title: Clinical Randomized Trial Investigating a Novel Pancreaticojejunostomy Technique for Pancreaticoduodenectomy in Patients With a High Risk for Postoperative Pancreatic Fistula
Brief Title: Evaluation of a Novel Pancreaticojejunostomy Technique for Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Christoph Ansorge, Christoph Ansorge, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKARV-GLH-001; KI-DSGE-DUAS (Other: Karolinska Institutet)
Record Dates: First submitted 2012-09-25; First posted 2012-10-02 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Pancreatic Fistula
Keywords: Postoperative pancreatic fistula; Pancreatic texture; Pancreatic duct diameter; Pancreatic consistency; Pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional anastomosis (No Intervention): Conventional anastomosis: The pancreaticojejunostomy is carried out in a traditional way according to "Cattell's duct-to-mucosa technique".
- Novel anastomosis (Active Comparator): Novel anastomosis: This the active comparator to the conventional anastomosis. A new pancreaticojejunostomy technique is used for the reconstruction. The pancreas is intubated into the jejunum.
  Interventions: Procedure: Pancreaticojejunostomy technique

INTERVENTIONS:
Procedure: Pancreaticojejunostomy technique — The anastomosis between jejunum and remnant pancreas has a pivotal impact on the incidence of postoperative pancreatic fistula. by this novel technique the remnant pancreas is intubated into the jejunum without extensive manipulation.
  Other Names: Pancreaticojejunal anastomosis; Intubating pancreaticojejunostomy; Dunking pancreaticojejunostomy; pancreatojejunostomy
  Arms: Novel anastomosis

SUMMARY:
Pancreaticoduodenectomy is a surgical procedure for removing cancer in the pancreas, the bile system or the duodenum that is associated with a high rate of complications. The study wants to investigate whether a new technique to reconstruct the joint between the pancreatic gland and the short bowel can reduce the rate of severe complications after this complex surgical procedure.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is a complex surgical procedure for radically resecting tumors in the pancreatic head, distal bile duct or duodenum. Postoperative pancreatic fistula is the main contributor of severe postoperative morbidity after pancreaticoduodenectomy. Characteristics of the pancreatic gland like soft pancreatic consistency and small pancreatic main duct predispose for the postoperative fistula development. In high risk patients, the risk of suffering from associated postoperative morbidity is 50 percent which is considered unacceptable high. The aim of the current trial is to investigate whether a new anastomosing technique for the pancreaticojejunostomy can reduce the incidence of associated postoperative morbidity in patients undergoing pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective pancreaticoduodenectomy
* Pancreatic gland with high risk criteria for associated postoperative morbidity

Exclusion Criteria:

* Patients do not accept participation
* Pancreatic gland with intermediate or low risk criteria for associated postoperative morbidity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2011-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Clinically Relevant Postoperative Pancreatic Fistula | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Postoperative pancreatic fistula as defined by the International Study Group of Pancreatic Fistula

SECONDARY OUTCOMES:
Associated postoperative morbidity | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Postoperative pancreatic fistula and abscesses or fluid collections adjacent to the pancreaticojejunostomy constitute a morbidity event; pancreaticojejunostomy-associated morbidity.

OTHER OUTCOMES:
Severity of postoperative complications | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The severity of postoperative complications as classified by the classification system of postoperative complications adopted for pancreatic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Ansorge, MD, PhD, Principal Investigator — Karolinska Institutet; Ralf Segersvärd, MD, PhD, Study Director — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Department of Upper Abdominal Surgery, Linköping University Hospital, Linköping
  - Department of Surgical gastroenterology, Karolinska University Hospital, Stockholm

REFERENCES:
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Ansorge C, Strommer L, Andren-Sandberg A, Lundell L, Herrington MK, Segersvard R. Structured intraoperative assessment of pancreatic gland characteristics in predicting complications after pancreaticoduodenectomy. Br J Surg. 2012 Aug;99(8):1076-82. doi: 10.1002/bjs.8784. Epub 2012 May 4. PMID 22556164
- [Background] Kennedy EP, Yeo CJ. Dunking pancreaticojejunostomy versus duct-to-mucosa anastomosis. J Hepatobiliary Pancreat Sci. 2011 Nov;18(6):769-74. doi: 10.1007/s00534-011-0429-y. PMID 21845376
- See also: Issuer organization — http://ki.se
- See also: Investigation site — http://www.karolinska.se
- See also: Investigation site — http://www.lio.se